CLINICAL TRIAL: NCT07054398
Title: Assessment of Serum Catestatin Level in Acne Vulgaris Patients Before and After Treatment With Oral Isotretinoin
Brief Title: Assessment of Serum Catestatin Level in Acne Vulgaris Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Mona Zakaria Mohamed, Resident of Dermatology, at Faculty of medicine, Aswan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Serum Catestatin
Record Dates: First submitted 2025-05-15; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin; chromogranin A (344-364)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Study Group) (Active Comparator): About 30 patients suffering from moderate and severe acne Vulgaris
  Interventions: Drug: Isotretinoin
- Group II (Control Group) (Placebo Comparator): About 30 Healthy persons
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — * Measure the serum levels of catestatin in patients with moderate and severe acne vulgaris versus healthy control persons.
  * Evaluate the effect of oral isotretinoin treatment on serum catestatin levels in patients with moderate and severe acne vulgaris.
  Other Names: Catestatin

SUMMARY:
Acne vulgaris is a persistent inflammatory condition of the pilosebaceous unit, affecting 85% of people between the ages of 12 and 24, it is regarded as one of the most common diseases in teenagers and young adults.

Catestatin, a peptide derived from chromogranin A (CgA), was first discovered in 1997 as an acute nicotinic-cholinergic antagonist. Later, it was determined that CST is a pleiotropic hormone.

DETAILED DESCRIPTION:
Acne vulgaris is a persistent inflammatory condition of the pilosebaceous unit, affecting 85% of people between the ages of 12 and 24, it is regarded as one of the most common diseases in teenagers and young adults.

Four factors are thought to be linked to the physiopathology of acne: changes in the keratinization process of corneocytes, which results in the development of comedones; follicular proliferation of the bacterium Cutibacterium acnes; increased production of inflammatory mediators, including interleukins (IL)-1β; and increased sebum production by the sebaceous gland.

The distinctive lesions can be classified as either inflammatory (papules, pustules, nodules, and cysts) or non-inflammatory (open/black and closed/white comedones). Both types of lesions cause skin pigmentation and scarring, which need consistent treatment. Lesions are usually found on the chest, upper back, neck, and face.

There are wide variety of topical and oral therapy methods can be used for acne treatment. Topical retinoids, benzoyl peroxide, azelaic acid, and their combinations are considered first-line agents. Oral drugs such as oral antibiotics, isotretinoin, or hormonal therapy may be used to treat refractory or more severe acne.

The most effective treatment for acne is still isotretinoin (13-cis-retinoic acid), an oral retinoid that was licensed in 1982 for the treatment of acne vulgaris. Multiple randomized controlled trials have confirmed that it is more effective than oral antibiotics and placebos at reducing the number of acne lesions.

Oral isotretinoin is the only medication that can cure or prolong remission of moderate to severe acne , avoiding scarring and psychological effects. isotretinoin reduces the size of sebaceous glands, lowers sebum excretion, regulates cell proliferation, decreases keratinization, and modifies the follicles' microenvironment , resulting in a decrease in the number of Cutibacterium acnes. Furthermore, it has immunomodulatory and anti-inflammatory qualities by lowering the expression of monocyte TLR-2, lowering the inflammatory cytokine response, and having anti-neoplastic effects.

Antimicrobial peptides (AMP) have a wide spectrum of antibacterial and immunomodulatory properties against bacteria (Gram positive and Gram negative), viruses and fungi.

Variations in AMP expression in the skin could play a significant role in the pathogenesis of numerous skin conditions, such as acne vulgaris.

Catestatin, a peptide derived from chromogranin A (CgA), was first discovered in 1997 as an acute nicotinic-cholinergic antagonist. Later, it was determined that CST is a pleiotropic hormone.

Catestatin (CST), a versatile 21 amino acid long cationic peptide, derived from the processing of chromogranin A, catestatin is produced by chromaffin cells and neutrophils , retained in chromaffin granules, and produced in the skin upon damage.

Catestatin affects innate immunity, inflammation, blood pressure regulation, and catecholamine inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons of both sexes with moderate and severe acne.

Exclusion Criteria:

* Pregnant and lactating women.
* Immunocompromised patients.
* Severe anemia.
* History of chronic liver disease.
* Hyperlipidemia
* Non-inflammatory acne conditions.
* History of neurologic disorders.
* History of neoplastic disorders.
* History of cardiac disease.
* History of systemic acne treatment for at least 4 weeks prior to inclusion and no topical treatments for at least 2 weeks.
* Cases with known hypersensitivity reaction to isotretinoin.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Evalaute serum level of Catestatin in acne patient | 12 weeks
  Assessment of clinical improvement according to:(8) G4(excellent:100% reduction) G3(good:75-99% reduction) G2(moderate: 50-74% reduction) G1(insufficient :1-49% reduction) G0(unchanged) G-1(worse)
Evalaute the effect of treatment with systemic isotretinon | 12 weeks
  Evaluate the effect of treatment with systemic isotretinon therapy (0.5 mg/kg/day, up to 40 mg daily) on the level of serum Catestatin on the Participants whom suffering from Acne Vulgaris whether moderate or severe.

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa Adam Ali El Taieb, Professor, Study Chair — Dermatology, Venereology and Andrology. Faculty of Medicine,Aswan University
Locations (1):
- Aswan Unuversity Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided